CLINICAL TRIAL: NCT06501326
Title: Clinical Efficacy and Safety of Liraglutide in the Treatment of Obesity Combined With Metabolism-associated Fatty Liver Disease (MAFLD)
Brief Title: Efficacy and Safety of Liraglutide in the Treatment of Obesity Combined With Metabolism Associated Fatty Liver Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: liraglutide
Record Dates: First submitted 2023-12-26; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-11

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Liraglutide; Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lifestyle intervention + orlistat group (Active Comparator): The control group was treated with lifestyle intervention + orlistat until the end of follow-up.
  Interventions: Drug: Orlistat
- lifestyle intervention + liraglutide group (Experimental): Trial group 1 was treated with lifestyle intervention + liraglutide.
  Interventions: Drug: Liraglutide
- lifestyle intervention + liraglutide + orlistat group (Experimental): Trial group 2 was treated with lifestyle intervention + liraglutide + orlistat for a total treatment and follow-up period of 3 months.
  Interventions: Drug: Liraglutide; Drug: Orlistat

INTERVENTIONS:
Drug: Liraglutide — After randomization, the control group was treated with lifestyle intervention + orlistat until the end of follow-up. Trial group 1 was treated with lifestyle intervention + liraglutide. Trial group 2 was treated with lifestyle intervention + liraglutide + orlistat for a total treatment and follow-up period of 3 months.
  Arms: lifestyle intervention + liraglutide + orlistat group; lifestyle intervention + liraglutide group
Drug: Orlistat — After randomization, the control group was treated with lifestyle intervention + orlistat until the end of follow-up. Trial group 1 was treated with lifestyle intervention + liraglutide. Trial group 2 was treated with lifestyle intervention + liraglutide + orlistat for a total treatment and follow-up period of 3 months.
  Arms: lifestyle intervention + liraglutide + orlistat group; lifestyle intervention + orlistat group

SUMMARY:
STUDY OBJECTIVE: To explore the clinical efficacy and safety of liraglutide in obesity combined with metabolism-associated fatty liver disease (MAFLD).

INTERVENTION PROGRAM: All subjects underwent dietary control and exercise therapy, and controlled smoking and alcohol consumption. During the 3 months of the trial, men were instructed to follow a diet of 1,500 to 1,800 kcal per day and women followed a diet of 1,200 to 1,500 kcal per day. All three diets included 40 to 55 percent carbohydrates, 15 to 20 percent protein and 20 to 30 percent fat. During the 3-month trial period, subjects performed at least 150 minutes of moderate-intensity exercise per week with an energy expenditure of 1500 kcal/week or more. Other medications containing the same ingredients as orlistat and liraglutide were prohibited during the trial period. After randomization, the control group was treated with lifestyle intervention + orlistat until the end of follow-up. Trial group 1 was treated with lifestyle intervention + liraglutide. Trial group 2 was treated with lifestyle intervention + liraglutide + orlistat for a total treatment and follow-up period of 3 months.

DETAILED DESCRIPTION:
1. Randomization Patients were divided into three groups by lifestyle intervention + orlistat treatment, in lifestyle intervention + liraglutide treatment and in lifestyle intervention + orlistat + liraglutide treatment, and eligible patients were randomized into trial group 1,2 and control group strictly according to the random number method. The ratio of test group 1,2 and control group was 1:1:1.
2. Name and specification of the intervention / study medication Use: liraglutide injection, 3ml: 18mg (prefilled pen) and orlistat capsules.
3. Study the intervention program All subjects were treated with dietary control and exercise therapy and controlled smoking and alcohol consumption.During the 3 months of the trial, men were instructed to follow a diet of 1500 to 1800 kcal per day and women followed a diet of 1200 to 1500 kcal per day. All three groups of diets included 40% to 55% carbohydrates, 15% to 20% protein and 20% to 30% fat.During the 3-month trial period, conduct at least 150 minutes of moderate intensity exercise per week, with exercise energy consumption of 1500 kcal / week or more.Other drugs containing the same ingredients of orlistat and liraglutide were prohibited during the trial.After randomization, the control group was treated with lifestyle intervention + orlistat until the end of follow-up.Trial Group 1 was treated with lifestyle intervention plus liraglutide.Trial Group 2 was treated with lifestyle intervention plus liraglutide plus orlistat.Medication regimen: Patients in the test or control groups were treated with liraglutide or (and) orlistat for 3 months from the first day after enrollment. The starting dose of liraglutide was 0.6mg per day, gradually increased to 1.2mg per day after one week, and continued to 1.8mg per day when tolerated. Patients taking orlistat should take 120mg orlistat capsules every day or one hour after a meal, and if one meal is not eaten or the food is not fat, they can be omitted.
4. Efficacy evaluation index (primary efficacy index and secondary efficacy index) glycosylated hemoglobin, FABP 4, body weight, waist circumference, hip circumference, BMI, and lipid index: TC, TG, HDL-C, LDL-C; Liver fibrosis index: liver hardness, liver fat attenuation (fibro scan detection instrument), body fat volume, visceral fat area (inbody body meter), liver function index: balanced and comparable analysis of ALT and AST before the treatment of the three groups of (1); (2) the change of each level before and after treatment, Test of their respective efficacy; (3) The difference between the three groups after treatment and the difference between the groups and the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Metabolic Associated Fatty Liver Disease(MAFLD);
2. Clinical diagnosis of Obesity.

Exclusion Criteria:

1. Medicated Hepatitis and Viral Hepatitis;
2. Have severe hepatic or renal insufficiency;
3. have used any weight-loss drug;
4. History of severe gastrointestinal disorders;
5. Malignant tumors, autoimmune diseases, hematologic diseases;
6. Psychopath;
7. Women who are pregnant, breastfeeding or preparing for pregnancy;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Body weight | Three months
  Body weight
FABP4 | Three months
  fatty acid-binding protein-4
BMI | Three months
  body mass index
lipid indices | Three months
  TC, TG, HDL-C, LDL-C
LSM | Three months
  liver stiffness measurement
CAP | Three months
  Controlled attenuation parameters

SECONDARY OUTCOMES:
Waist circumference, | Three months
  Waist circumference
hip circumference | Three months
  hip circumference

CONTACTS AND LOCATIONS:
Overall Officials: GU Yunjuan, doctor, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No